CLINICAL TRIAL: NCT06602453
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of GDC-8264 in Preventing Cardiac Surgery-Associated Acute Kidney Injury and Major Adverse Kidney Events
Brief Title: A Study to Evaluate the Efficacy and Safety of GDC-8264 in Preventing Cardiac Surgery-Associated Acute Kidney Injury (AKI) and Major Adverse Kidney Events (MAKE)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC45428; 2024-513125-23-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: GDC-8264 (Experimental): Participants will receive GDC-8264 as per a pre-defined dosing regimen in Part 1.
  Interventions: Drug: GDC-8264
- Part 1: Placebo (Placebo Comparator): Participants will receive GDC-8264 matching placebo as per a pre-defined dosing regimen in Part 1.
  Interventions: Drug: Placebo
- Part 2: GDC-8264 (Experimental): Participants will receive GDC-8264 as per a pre-defined dosing regimen in Part 2.
  Interventions: Drug: GDC-8264
- Part 2: Placebo (Placebo Comparator): Participants will receive GDC-8264 matching placebo as per a pre-defined dosing regimen in Part 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GDC-8264 — GDC-8264 will be administered as per pre-defined regimen.
  Other Names: RO7288817
  Arms: Part 1: GDC-8264; Part 2: GDC-8264
Drug: Placebo — Placebo will be administered as per pre-defined regimen.
  Arms: Part 1: Placebo; Part 2: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of GDC-8264 compared with placebo in participants undergoing cardiac surgery who are determined to be at moderate to high risk of developing AKI and subsequent MAKE at 90 days after surgery (MAKE90). The study will be performed in two parts- Part 1 and Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. One of the following non-emergent cardiac surgery types that requires cardiopulmonary bypass (CPB) to be done in one procedure rather than separate procedures: Isolated Coronary Artery Bypass Grafting (CABG); Isolated Surgical Aortic Valve Replacement (AVR), Mitral Valve Replacement (MVR), Mitral Valve repair (MVr); Combined CABG+AVR, CABG+MVR, CABG+MVr, AVR+MVR, AVR+MVr
2. At least one or at least two of the following AKI risk factors, depending on the type of surgery: age > 70 years, history of CKD with eGFR < 60 milliliters/ minutes/ 1.73 meter square (ml/min/1.73 m^2) within the last 6 months, diabetes (type 1 or type 2) requiring at least one oral hypoglycemic agent or insulin, history of chronic obstructive pulmonary disease (COPD) requiring medical therapy, left ventricular ejection fraction (LVEF) < 40%, preoperative anemia [hemoglobin <10 grams/deciliters (g/dL)]
3. Stable kidney function with no known episodes of AKI within 2 weeks of screening

Exclusion Criteria:

1. Need for renal replacement therapy (peritoneal dialysis or hemodialysis)
2. Need for intra-aortic balloon pump, temporary mechanical circulatory support, or extracorporeal membrane oxygenation prior to scheduled surgery
3. Presence of a durable left ventricular assist device
4. Need for concurrent aortic surgery that requires circulatory arrest and deep hypothermia or repair of congenital heart defects
5. Heart transplant
6. Transcatheter valve replacements
7. Hypotension or shock requiring hospital admission
8. Cardiopulmonary resuscitation
9. eGFR < 20 mL/min/1.73 m^2
10. Heart failure with ejection fraction < 20%, or episode of decompensated heart failure requiring intervention within 2 weeks prior to screening
11. History of kidney transplant or only one kidney (due to donation)
12. Renal agenesis, total nephrectomy, or partial nephrectomy of > 50%

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Develop MAKE90 | From Day 0 (day of surgery) up to Day 90 post-surgery
Number of Participants With Adverse Events (AEs) | Up to Day 90 post surgery

SECONDARY OUTCOMES:
Percentage of Participants who Develop AKI | From Day 0 (day of surgery) up to Day 7 post surgery
Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline up to Days 30, 60 and 90 post surgery
Number of Participants With New or Worsened Chronic Kidney Disease (CKD) | Baseline up to Day 90 post surgery
Percentage of Participants who Develop MAKE30 and MAKE60 | From Day 0 (day of surgery) to Day 30, Day 60 post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- United States (16):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of Stanford Medical Center, Stanford, California
  - Yale School of Medicine Yale New Haven Hospital, New Haven, Connecticut
  - James A Haley Veteran Affairs Medical Center - NAVREF - PPDS, Tampa, Florida
  - John Hopkins Hospital, Lutherville, Maryland
  - Baystate Cardiac Surgery, Springfield, Massachusetts
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - CHI Health Nebraska Heart, Lincoln, Nebraska
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Wake Forest University School of Medicine - PPDS, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Richmond VA Medical Center NAVREF PPDS, Richmond, Virginia
  - Aurora St Lukes Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - Gold Coast University Hospital, Southport, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - ZOL Genk campus Sint Jan, Genk
  - UZ Leuven, Leuven
  - Hopital de la Citadelle, Liège
- Saint John Regional Hospital, Saint John, New Brunswick, Canada
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
- France (3):
  - CHU Angers, Angers
  - APHP - Hopital de la Pitie Salpetriere, Paris
  - CHU de Reims, Reims
- Germany (2):
  - Herzzentrum Dresden GmbH Universitatsklinikum, Dresden
  - Universitätsklinikum Essen, Essen
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
- South Korea (2):
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
- Spain (4):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Universitario de La Princesa, Madrid
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing